CLINICAL TRIAL: NCT01246141
Title: The Institute of Cardiovascular Surgery
Brief Title: The Comparison of Tricuspid Replacement and Repair in Patients With Combined Heart Valve Disease
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: zhang jinzhou, the departement of cardiovascular surgery, xijing hospital
Other Study IDs: 20101012
Record Dates: First submitted 2010-11-20; First posted 2010-11-23 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 1998-01

CONDITIONS: Tricuspid Valve Regurgitation
Keywords: tricuspid valve regurgitation; replacement; repair; outcomes
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Repair group: patients in repair group underwent tricuspid repair for functional tricuspid regurgitation.
- replacement group: In this group, patients underwent tricuspid valve replacement for functional tricuspid regurgitation.

SUMMARY:
Functional tricuspid regurgitation is common in patients with heart valve disease, replacement and repair both can correct this anomaly. However, there is no data to address which one can bring more benefits to these patients with combined heart valve disease. The investigators retrospectively review patients with two or more heart valve disease and functional tricuspid regurgitation, and assess its long term outcomes.

DETAILED DESCRIPTION:
we reviewed patients who admitted to our hospital due to combined heart valve disease, and underwent tricuspid valve replacement or repair from January,1998 to december,2009. we made a comparison between these two groups, in term of early results after operation and long term results.

ELIGIBILITY:
Inclusion Criteria:

* Significant disorders in aortic and mitral valves
* Moderate ～ severe tricuspid regurgitation
* Underwent tricuspid repair or replacement operation

Exclusion Criteria:

* Isolate tricuspid valve lesion
* Mild tricuspid valve regurgitation
* Tricuspid valve regurgitation was left without surgical treatment

Ages: 21 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with aortic valve and mitral valve diseases and functional tricuspid valve regurgitation underwent surgical operations from Nov., 1998 to Dec., 2009 in our institute.
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 1998-01; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: zhang jinzhou, MD, Principal Investigator — Xijing Hospital
Locations (1):
- Zhang Jinzhou, Xi'an, Shaanxi, China